CLINICAL TRIAL: NCT02759562
Title: A Phase 2b, Dose-Ranging Study of the Effect of GS-5745 on FEV1 in Adult Subjects With Cystic Fibrosis
Brief Title: Effect of Andecaliximab on FEV1 in Adults With Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of development for this indication
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-404-1808; 2015-002192-23 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — andecaliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Andecaliximab 600 mg (Part 1) (Experimental): Andecaliximab 600 mg weekly for 8 weeks
  Interventions: Drug: Andecaliximab
- Placebo (Part 1) (Placebo Comparator): Placebo weekly for 8 weeks
  Interventions: Drug: Placebo
- Andecaliximab 300 mg (Part 2) (Experimental): Andecaliximab 300 mg weekly for 8 weeks
  Interventions: Drug: Andecaliximab
- Andecaliximab 150 mg (Part 2) (Experimental): Andecaliximab 150 mg + placebo weekly for 8 weeks
  Interventions: Drug: Andecaliximab; Drug: Placebo
- Placebo (Part 2) (Placebo Comparator): Placebo weekly for 8 weeks
  Interventions: Drug: Placebo
- Open-Label Extension (Experimental): (Part 1) Andecaliximab 600 mg weekly for 16 weeks; (Part 2) Andecaliximab 300 mg weekly for 16 weeks
  Interventions: Drug: Andecaliximab

INTERVENTIONS:
Drug: Andecaliximab — Administered via subcutaneous injection
  Other Names: GS-5745
  Arms: Andecaliximab 150 mg (Part 2); Andecaliximab 300 mg (Part 2); Andecaliximab 600 mg (Part 1); Open-Label Extension
Drug: Placebo — Administered via subcutaneous injection
  Arms: Andecaliximab 150 mg (Part 2); Placebo (Part 1); Placebo (Part 2)

SUMMARY:
The primary objective of this study is to evaluate the effect of andecaliximab (GS-5745) on pre-bronchodilator forced expiratory volume in 1 second (FEV1) % predicted in adults with cystic fibrosis (CF) after 8 weeks of treatment.

There will be 2 parts to this study. In Part 1, andecaliximab 600 mg or placebo will be administered for 8 weeks. In Part 2, andecaliximab 300 mg, 150 mg, or placebo will be administered for 8 weeks. Part 2 will be initiated after completion of Part 1.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of CF as determined by the 2008 Cystic Fibrosis Foundation Consensus Report criteria
* Must have a body weight of > 40 kg (88.2 lb) at study screening
* Pre-bronchodilator FEV1 ≥ 40% and ≤ 80% of predicted at screening
* Two pre-bronchodilator spirometry measures during screening and baseline must meet the following 2 criteria:

  * The relative difference of FEV1(L), calculated as the absolute value of [(first FEV1 - second FEV1) / first FEV1] x 100 should be < 12% AND
  * The absolute difference in FEV1 should be < 200 ml
* Negative Sputum Investigation/History of any Mycobacterium spp. or Burkholderia spp. per specified protocol-defined time periods
* Clinically stable with no evidence of significant respiratory symptoms that would require administration of IV antibiotics, oxygen supplementation, or hospitalization within 30 days of baseline.
* On stable CF chronic medical regimen for at least 30 days prior to baseline and expected to remain stable through the completion of the study. This includes but is not limited to: chronic azithromycin use, inhaled bronchodilators, inhaled corticosteroids, inhaled dornase alpha, inhaled hypertonic saline, inhaled mannitol, ivacaftor, and/or ivacaftor/lumacaftor.

Key Exclusion Criteria:

* Concurrent use of oral antibiotics (excluding chronic azithromycin use) or IV antibiotics within 30 days of baseline. Prophylactic and chronic doxycycline use is prohibited during the study.
* Hospitalization for a respiratory event within 30 days of baseline
* Current use of systemic immunosuppressive drugs including oral corticosteroids within 30 days of Baseline
* Current requirement for daily continuous oxygen supplementation or requirement (medically necessary) of more than 2 L/minute at night (subject would not meet this exclusion criterion if supplemental oxygen is used for comfort only)
* History of solid organ (including lung) or hematologic transplant, or currently on a transplant waiting list

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- New Lambton, New South Wales, Australia
- Montpellier, France
- Berlin, Germany
- Barcelona, Spain
- Liverpool, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia and Europe. The first participant was screened on 04 November 2016. The last study visit occurred on 21 July 2017. The study was terminated after 6 participants were enrolled in Part 1 of the study. Therefore, Part 2 was not initiated.
Pre-assignment Details: 26 participants were screened.
Groups:
- Andecaliximab: Double-Blind Period: Andecaliximab 600 mg administered via subcutaneous injection weekly for 8 weeks
  Open-Label Period: Andecaliximab 600 mg administered via subcutaneous injection weekly for up to 16 weeks
- Placebo: Double-Blind Period: Placebo administered via subcutaneous injection weekly for 8 doses
  Open-Label Period: Andecaliximab 600 mg administered via subcutaneous injection weekly for up to 16 weeks
Period: Double-Blind Treatment Period (8 Weeks)
Arm/Group | Andecaliximab | Placebo
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Open-Label Treatment Period
Arm/Group | Andecaliximab | Placebo
Started (2 participants completed the Double-Blind Phase, but did not enter in the Open-Label Phase.) | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Withdrew Consent | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Andecaliximab | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (20.42) | 43.3 (10.02) | 44.7 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 1 | 1 | 2
  Australia | 1 | 0 | 1
  France | 0 | 1 | 1
  Germany | 0 | 1 | 1
  Spain | 1 | 0 | 1
Pre-bronchodilator Forced expiratory volume in 1 second (FEV1) % predicted [Mean (Standard Deviation); unit: percent] — FEV1 % predicted is defined as FEV1 of the patient divided by the average FEV1 in the population for any person of similar age, sex, race, and body composition.
  percent | 49.7 (8.70) | 59.1 (19.26) | 54.4 (14.33)
Post-bronchodilator FEV1 % predicted [Mean (Standard Deviation); unit: percent] | 52.1 (5.90) | 64.6 (20.58) | 58.3 (15.17)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Pre-bronchodilator FEV1 Percent Predicted From Baseline to Week 8
Time Frame: Baseline; Week 8
Population: Full Analysis Set: all randomized participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Andecaliximab | Placebo
Number analyzed (Participants) | 3 | 3
percent | -2.10 (4.446) | 2.90 (3.461)

2. Secondary Outcome: Absolute Change in Post-bronchodilator FEV1 Percent Predicted From Baseline to Week 8
Time Frame: Baseline; Week 8
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Andecaliximab | Placebo
Number analyzed (Participants) | 3 | 3
percent | 1.01 (4.534) | -1.45 (1.655)

3. Secondary Outcome: Relative Change in Pre-bronchodilator FEV1 Percent Predicted From Baseline to Week 8
Time Frame: Baseline; Week 8
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Andecaliximab | Placebo
Number analyzed (Participants) | 3 | 3
percent change | -3.85 (9.009) | 4.41 (4.196)

4. Secondary Outcome: Relative Change in Post-bronchodilator FEV1 Percent Predicted From Baseline to Week 8
Time Frame: Baseline; Week 8
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Andecaliximab | Placebo
Number analyzed (Participants) | 3 | 3
percent change | 2.28 (9.323) | -1.98 (1.749)

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure: 140 days)
Description: Safety Analysis Set
Groups:
- Andecaliximab (Double-Blind): Andecaliximab 600 mg administered via subcutaneous injection weekly for 8 weeks
- Placebo (Double-Blind): Placebo administered via subcutaneous injection weekly for 8 doses
- Andecaliximab (Open-Label): Andecaliximab 600 mg administered via subcutaneous injection weekly for up to 16 weeks
Arm/Group | Andecaliximab (Double-Blind) | Placebo (Double-Blind) | Andecaliximab (Open-Label)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab (Double-Blind) (N=3) | Placebo (Double-Blind) (N=3) | Andecaliximab (Open-Label) (N=4)
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 0 | 0
Injection site pruritus (General disorders) | 1 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Bacterial test positive (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Gilead made a decision to discontinue the development of andecaliximab in cystic fibrosis. This decision was not due to any safety concerns. Because only 6 participants were enrolled, no inferential analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT02759562/Prot_000.pdf
  • Study Protocol: Amendment 2 (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02759562/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT02759562/SAP_002.pdf